CLINICAL TRIAL: NCT05635084
Title: A First-in-human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenously Administered YN001 in Healthy Subjects
Brief Title: A First-in-human Study of YN001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YN001-001
Record Dates: First submitted 2022-10-20; First posted 2022-12-02 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YN001 (Experimental): YN001 (with a strength of 5 mL:10 mg). Subjects will be administered 250 to 500 mL of YN001 diluted in 5% dextrose injection up to 120 min(which allows a +/-5 min infusion window) intravenous infusion.
  Interventions: Drug: YN001
- Matching placebo for YN001 (Placebo Comparator): Matching placebo for YN001 is 5% dextrose injection. Subjects will be administered 250 to 500mL of 5% dextrose injection up to 120 min (which allows a +/-5 min infusion window) intravenous infusion.
  Interventions: Drug: Placebo for YN001

INTERVENTIONS:
Drug: YN001 — Dose ranges from 2-90mg
  Arms: YN001
Drug: Placebo for YN001 — 5% dextrose injection to mimic the YN001
  Other Names: YN001
  Arms: Matching placebo for YN001

SUMMARY:
This will be a single center, randomized, double-blind, placebo-controlled, single ascending dose and multiple ascending dose study in healthy adult subjects.

DETAILED DESCRIPTION:
A total of approximately 73 to 89 healthy male and female subjects will be enrolled into this study, it includes two parts:

Part A is single ascending dose stage, approximately 49 to 65 healthy subjects will be enrolled into about eight to ten cohorts. Subjects who meet eligibility criteria at screening will be admitted for baseline evaluations (Day -1). All baseline safety evaluation results must be available prior to dosing. The doses will be progressively escalated, with a sentinel dosing strategy employed for all cohorts.

Part B is multiple ascending dose stage, approximately 24 healthy subjects will be enrolled into about three cohorts. Subjects who meet eligibility criteria at screening will be admitted for baseline evaluations (Day -1). All baseline safety evaluation results must be available prior to dosing. The cohort M1 will be initiated by decision of SRC(safety review committee), then the doses will be progressively escalated.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Healthy male and female adults aged from 18 to 55 Years of age included, and in good health as determined by past medical history, physical examination, and vital signs, electrocardiogram, and laboratory tests at screening.
3. At screening, and baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for at least three (3) minutes.
4. Weigh at least 50 kg, and have a body mass index (BMI) within the rage of 18-32 kg/m2.
5. Willing and able to comply with the requirements of the study.

Exclusion Criteria:

Subjects fulfilling any of the following criteria are not eligible for inclusion in this study.

1. Receiving an investigational agent at the time of enrollment, or within 30 days or 5 half-lifes of enrollment, whichever is longer prior to study drug administration.
2. Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, COVID-19 vaccine, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing. If needed, (i.e., an incidental and limited need of maximum 2 g per day, no more than 3 consecutive days within 2 weeks prior to dosing) paracetamol is acceptable, but must be documented in the Concomitant medications page of the CRF.
3. Fasting triglyceride concentration >2.8 mmol/L.
4. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at Screening or Baseline:

   * PR > 220 msec
   * QRS complex > 120 msec
   * QTcB > 450 msec (males)
   * QTcB > 470 msec (females)
5. Pregnant or nursing (lactating) women.
6. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant UNLESS the subject agrees to comply with highly effective, double barrier contraception for the entire duration of the study and for a period of 30 days after the dose of study drug. Fertile males, defined as all males physiologically capable of conceiving offspring UNLESS the subject agrees to comply with highly effective, double barrier contraception for the entire duration of the study and for a period of 30 days after the dose of study drug.
7. Smokers (use of tobacco products in the previous 1 month). Urine cotinine levels will be measured during screening and at baseline for all subjects. Smokers will be defined as any subject who reports tobacco use and/or who has a urine cotinine ≥ 500 ng/mL. For light smokers to pass the cotinine test, smoking should be stopped at least 24 hours prior to reporting to the center (i.e., Day -2, early morning). Smoking will not be allowed during the study.
8. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays for alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates conducted during screening and/or baseline. Any THC-containing products should not be used at least 7 days prior to screening, and participant needs to abstain any THC-containing products during the trial. Alcohol abuse was defined as consumption of 14 or more standard drinks per week.
9. A positive hepatitis B surface antigen (HBsAg), or positive hepatitis C virus (HCV) or human immunodeficiency virus (HIV) test result.
10. A positive COVID-19 test result.
11. History of myopathy/myalgia, or susceptible to myopathy/rhabdomyolysis (e.g., hypothyroidism, family history of hereditary myopathy, previous muscle toxicity with HMG-CoA reductase inhibitors or fibrates).
12. Multiple drug allergies, or history of allergic reactions to rosuvastatin or any components of the study drug.
13. Donation or loss of more than 400 mL of blood within 3 months prior to study drug administration.
14. Plasma donation (> 100 ml) within 60 days prior to first dosing.
15. Hemoglobin levels below 12.0 g/dl at screening.
16. Recent (within the last 3 years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
17. Recent (within the last 3 years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated), or cardiac dysfunction or myocardial infarction.
18. History of significant food allergies (e.g. anaphylactic reactions). Mild (non-anaphylactic, hypersensitivity) food allergies such as lactose intolerance/glucose intolerance are permitted.
19. Any surgical or medical condition which might significantly alter the distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:

    * Inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding in the last 6 months;
    * Pancreatic injury or pancreatitis in the last 6 months;
    * Liver disease or liver injury as indicated by abnormal liver function tests such as SGOT (AST), SGPT (ALT), γ-GT, alkaline phosphatase, or serum bilirubin. The Investigator should be guided by the following criteria:
    * Any single parameter of ALT, AST, γ-GT, alkaline phosphatase, or serum bilirubin must not exceed 1.5 x upper limit of normal (ULN).
    * Any elevation above ULN of more than one parameter of ALT, AST, γ-GT, alkaline phosphatase, or serum bilirubin excludes a subject from participation in the study.

    If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to randomization, to rule out any laboratory error.
    * History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or BUN and/or urea values, or abnormal urinary constituents (e.g., albuminuria).
    * Evidence of urinary obstruction or difficulty in voiding at screening.
20. Significant illness resolved within two (2) weeks prior to initial dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of intravenously administered YN001 in healthy subjects. | Up to 15 days of last dose
  To evaluate the incidence of Adverse Events as Assessed by CTCAE v5.0, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities, Clinically Significant Physical Examination Abnormalities and Infusion Reaction.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the collection time point of the last measurable concentration (AUC0-t) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Area under the plasma concentration-time curve to infinity(AUCinf) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Maximum plasma concentration(Cmax) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Time of maximum concentration (Tmax) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Clearance(CL) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Elimination half-life (t1/2) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Volume of distribution estimates (Vdss) | Up to 168 hours of post initiation of last dose
  To evaluate the pharmacokinetics (PK) characteristics of of intravenously administered YN001 in healthy subjects.
Immunogenicity | Up to 168 hours of post initiation of last dose
  To evaluate the immunogenicity YN001 in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gonen, Ph.D, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No